CLINICAL TRIAL: NCT02076711
Title: Myocardial Efficiency of the Left Ventricle in Asymptomatic Patients With Aortic Valve Stenosis - a Prognostic Marker and a Target for Intervention?
Acronym: MELVAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Wiggers, Senior consultant, Assoc. professor, DMSc, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201300114731
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Aortic Stenosis
Keywords: Aortic Stenosis; Myocardial efficiency
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): Metoprololsuccinate
  Interventions: Drug: Metoprololsuccinate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoprololsuccinate
  Arms: Active
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Background - Aortic valve stenosis (AS) is the most common heart valve disease among adults in the Western world with a prevalence of 3 % in people older than 75 years of age. AS usually deteriorates over time leading to heart failure, with high mortality if aortic valve replacement (AVR) is not performed. Thus optimal timing of AVR is crucial, but can be challenging. Increasing life expectancy in our society will augment the therapeutic and socio economic impact of AS disease on our health care system. Therefore, new techniques for monitoring asymptomatic AS patients are needed. A potential approach is monitoring of LV myocardial efficiency (mechanical work/oxygen consumption). These measures have been suggested to be involved in the progression of non-valvular heart failure and closely related to prognosis, but never applied in a larger population of patients with AS. At present there are no recognized pharmacological treatments of AS. It is known that beta-blocker treatment in non-valvular systolic heart failure reduce heart rate, improves LV myocardial efficiency and reduces mortality. However, in patients with AS, the effects of beta-blockers are unknown.

Hypotheses - Treatment with the beta-blocker metoprolol succinate in patients with asymptomatic moderate to severe AS has beneficial effects on LV myocardial oxidative metabolism, myocardial efficiency and contractile function.

Objectives - To investigate if beta-blocker treatment in patients with moderate to severe, asymptomatic AS has beneficial effects on LV myocardial efficiency, contractile function and physical performance.

Design - A randomized double blind placebo controlled intervention trial. 40 patients with asymptomatic AS will be randomized to either per oral metoprolol succinate (N = 20) or placebo (N= 20) for 22 weeks.

Primary objective - Changes in myocardial efficiency

Secondary objectives - Myocardial oxygen consumption, Myocardial perfusion at rest, LV myocardial function, LVmass, Aortic valve area and transaortic valve velocities, 6 minute walking distance, N-terminal prohormone of brain natriuretic peptide, Quality of life (estimated by Minnesota living with heart failure questionnaire), LV wall stress

Methods - Patients will undergo echocardiography (resting and exercise), [11C]acetate PET and cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve area ≤1,2 cm2 and/or transaortic maximal velocity (VmaxAO) of 3,0-5,0 m/s
* Sinus rhythm >60/min after 5 minutes of rest
* LVEF >≥50%
* Male or female
* Age 20-100 years old
* Safe birth control management for women of childbearing potential.
* Negative urine-HCG for women of childbearing potential
* Ability to understand the written patient information and to give informed consent

Exclusion Criteria:

* Systolic BP <100 mmHg after 5 minutes of rest
* Left ventricular posterior wall thickness >17 mm
* Signs or history of major myocardial infarction and/or severe ischemic heart disease
* Severe asthma or chronic obstructive pulmonary disease
* New York Heart Association (NYHA) classification > I due to AS
* NYHA > II due to non-cardiac causes
* 2ᵒ or 3ᵒ atrioventricular block
* Ongoing beta-blocker therapy
* Ongoing verapamil or diltiazem therapy
* Ongoing monoamine oxidase inhibitors therapy (except MAO-B-inhibitors)
* Sick sinus syndrome
* Atrial fibrillation or fluttering
* Lack of stable sinus rhythm
* Pheochromocytoma
* Severe peripheral vascular disease
* Intolerance of Metoprolol succinate or its excipients
* Other disease or treatment making subject unsuitable for study participation
* Intolerance of tracer used for [11C]acetate PET recordings
* Participation in other intervention study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
LV myocardial efficiency | Changes will be evaluated after an expected average of 22 weeks of treatment

SECONDARY OUTCOMES:
LV oxygen consumption | Changes will be evaluated after an expected average of 22 weeks of treatment
LV perfusion | Changes will be evaluated after an expected average of 22 weeks of treatment
LV myocardial function | Changes will be evaluated after an expected average of 22 weeks of treatment
LVmass | Changes will be evaluated after an expected average of 22 weeks of treatment
Aortic valve area | Changes will be evaluated after an expected average of 22 weeks of treatment
Transaortic valve velocities | Changes will be evaluated after an expected average of 22 weeks of treatment
6 minute walking distance | Changes will be evaluated after an expected average of 22 weeks of treatment
N-terminal prohormone of brain natriuretic peptide | Changes will be evaluated after an expected average of 22 weeks of treatment
Quality of life - estimated by Minnesota living with heart failure questionnaire | Changes will be evaluated after an expected average of 22 weeks of treatment
LV wall stress | Changes will be evaluated after an expected average of 22 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Wiggers, DMSc, Principal Investigator
Locations (1):
- Aarhus University Hospital, Department of Cardiology, Brendstrupgaardsvej 100, Aarhus N, Denmark

REFERENCES:
- [Derived] Hansson NH, Sorensen J, Harms HJ, Kim WY, Nielsen R, Tolbod LP, Frokiaer J, Bouchelouche K, Dodt KK, Sihm I, Poulsen SH, Wiggers H. Metoprolol Reduces Hemodynamic and Metabolic Overload in Asymptomatic Aortic Valve Stenosis Patients: A Randomized Trial. Circ Cardiovasc Imaging. 2017 Oct;10(10):e006557. doi: 10.1161/CIRCIMAGING.117.006557. PMID 28956773